CLINICAL TRIAL: NCT03580928
Title: A Phase 2 Study of Acalabrutinib, Venetoclax, and Obinutuzumab (AVO) for Initial Therapy of Chronic Lymphocytic Leukemia
Brief Title: Acalabrutinib, Venetoclax, and Obinutuzumab for Initial Therapy of CLL
Acronym: AVO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: AstraZeneca (Industry); Genentech, Inc. (Industry); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Matthew S. Davids, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-226; 1R01CA266298-01A1 (NIH)
Record Dates: First submitted 2018-06-25; First posted 2018-07-10 (Actual); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
Keywords: Chronic Lymphocytic Leukemia (CLL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — venetoclax; obinutuzumab; acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Acalabrutinib/Venetoclax/Obinutuzumab (AVO) with non-high-risk CLL disease (Experimental): * Acalabrutinib will be administered orally twice daily at 100 mg bid
  * Venetoclax will be administered orally once daily, with dose ramp-up from 20 mg up to a final dose of 400 mg
  * Obinutuzumab will be administered as per standard of care for 6 months with dosing at 100 mg on cycle 1 day 1, 900 mg on cycle 1 day 2, and then 1,000 mg on cycle 1 days 8, 15, and day 1 of cycles 2-6
  Interventions: Drug: Venetoclax; Drug: Obinutuzumab; Drug: Acalabrutinib
- Acalabrutinib/Venetoclax/Obinutuzumab (AVO) with high-risk CLL disease (Experimental): * Acalabrutinib will be administered orally twice daily at 100 mg bid
  * Venetoclax will be administered orally once daily, with dose ramp-up from 20 mg up to a final dose of 400 mg
  * Obinutuzumab will be administered as per standard of care for 6 months with dosing at 100 mg on cycle 1 day 1, 900 mg on cycle 1 day 2, and then 1,000 mg on cycle 1 days 8, 15, and day 1 of cycles 2-6.
  High-risk CLL disease (cohort 2), defined as 17p deletion and/or TP53 mutation
  Interventions: Drug: Venetoclax; Drug: Obinutuzumab; Drug: Acalabrutinib

INTERVENTIONS:
Drug: Venetoclax — Venetoclax is an oral drug that blocks the function of a protein called BCL-2. CLL cancer cells are thought to depend on the BCL-2 protein for their survival. By blocking BCL-2, venetoclax may kill cancer cells or stop them from growing.
  Other Names: Venclexta
Drug: Obinutuzumab — Obinutuzumab is a type of drug called a monoclonal antibody. It targets a protein CD20 on the surface of the CLL cell, causing it to die
  Other Names: Gazyva
Drug: Acalabrutinib — Acalabrutinib is a type of drug called a kinase inhibitor. It blocks a type of protein called Bruton Tyrosine Kinase (BTK) that helps CLL cells live and grow
  Other Names: Calquence

SUMMARY:
This research study is evaluating the combination of three drugs - acalabrutinib, venetoclax, and obinutuzumab -- as a possible treatment for chronic lymphocytic leukemia (CLL).

The drugs involved in this study are:

* Acalabrutinib
* Venetoclax
* Obinutuzmab

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of investigational drugs to learn whether the drugs work in treating a specific disease. "Investigational" means that the drugs are being studied. The FDA (the U.S. Food and Drug Administration) has not approved acalabrutinib for CLL, although it is FDA-approved for patients with relapsed mantle cell lymphoma. The FDA has approved venetoclax and obinutuzumab separately for the treatment of patients with CLL. However, the FDA has not approved the combination of these three drugs together (acalabrutinb, venetoclax, and obinutuzumab) as a treatment for any disease. This combination is investigational. In this research study, the investigators are trying to learn if giving the three drugs together can safely and effectively treat CLL.

Acalabrutinib is a type of drug called a kinase inhibitor. It blocks a type of protein called Bruton Tyrosine Kinase (BTK) that helps CLL cells live and grow. By blocking BTK, acalabrutinib may kill cancer cells or stop them from growing. As of September 2017, acalabrutinib has been administered to more than 2,000 people including healthy volunteers, patients with cancers, and patients with rheumatoid arthritis. A few hundred patients with CLL have been treated with acalabrutinib as a single drug, and some of these patients had improvement of their cancer with this treatment.

Obinutuzumab is a type of drug called a monoclonal antibody. It targets a protein on the surface of the CLL cell, causing it to die. Obintuzumab has already been shown to be safe and effective at treating CLL, and is FDA-approved when given together with chemotherapy.

Venetoclax is an oral drug that blocks the function of a protein called BCL-2. CLL cancer cells are thought to depend on the BCL-2 protein for their survival. By blocking BCL-2, venetoclax may kill cancer cells or stop them from growing. Venetoclax has been shown to be safe and effective when given alone to treat patients with CLL and is FDA-approved for patients with CLL after their disease has worsened after at least 1 prior therapy.

If, after 15 or 24 cycles of this investigational therapy, participants have a complete response to the drugs in this trial -- meaning that the investigators cannot detect any CLL using CT scans, bone marrow biopsy and a sensitive test called minimal residual disease (MRD) testing -- participants will stop therapy with acalabrutinib and venetoclax. The investigators will continue to monitor participants while they are off of therapy, and if the CLL comes back participants will be able to restart acalabrutinib and venetoclax. The use of MRD testing to identify small amounts of CLL is investigational, meaning that it has not been FDA-approved. The use of results from this test to guide the decision to stop and re-start therapy, as is done in the trial here, is also investigational.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have CLL or SLL
* In cohort 2, subjects must have TP53-aberrant disease defined as:

  * Del(17p) detected on karyotype and/or FISH; OR
  * TP53 mutation
* Participants must have measurable disease (lymphocytosis > 5,000 / µl, or palpable or CT measurable lymphadenopathy ≥ 1.5 cm, or bone marrow involvement ≥30%).
* Subjects must not have received any prior systemic therapy for CLL or SLL due to meeting IWCLL 2018 guidelines and must currently have an indication for treatment as defined by the IWCLL 2018 guidelines:

  * Massive or progressive or symptomatic splenomegaly; OR
  * Massive lymph nodes, nodal clusters, or progressive lymphadenopathy; OR
  * Significant fatigue (i.e. ECOG PS 2 or worse; cannot work or unable to perform usual activities); OR
  * Fever ≥ 100.5°F for 2 or more weeks without evidence of infection; OR
  * Night sweats for ≥ 1 months without evidence of infection; OR
  * Presence of weight loss ≥ 10% over the preceding 6 months; OR
  * Progressive lymphocytosis with an increase of ≥ 50% over a 2-month period or lymphocyte doubling time of less than 6 months; OR
  * Evidence of progressive marrow failure as manifested by the development of or worsening of anemia and/or thrombocytopenia; OR
  * Autoimmune anemia and/or thrombocytopenia that is poorly responsive to corticosteroids and another standard therapy such as rituximab; OR
  * Symptomatic or functional extranodal involvement
* Age greater than or equal to 18 years.
* ECOG performance status ≤2
* Participants must have adequate organ and marrow function as defined below:

  * total bilirubin ≤1.5 times upper limit of normal, unless there is disease involvement of the liver, hemolysis, or a known history of Gilbert's disease, in which case direct bilirubin must be ≤3 times the upper limit of normal
  * AST and ALT ≤ 2.5 times the upper limit of normal. If there is hemolysis or documented disease involvement of the liver, then patients with any AST or ALT abnormalities remain eligible.
  * creatinine clearance (CrCl) ≥ 50 mL/min using 24-hour urine collection for creatinine clearance or calculated CrCl
  * PT/INR ≤2 times the upper limit of normal and PTT ≤2 times the upper limit of normal
  * Absolute neutrophil count ≥750 cells/mm3 or ≥500 cells/mm3 in subjects with documented bone marrow involvement
  * Platelet count without transfusional support must be ≥50,000 cells/mm3 or ≥ 30,000 cells/mm3 in subjects with documented bone marrow involvement
* Pregnant or lactating

Exclusion Criteria:

* Participants who have a history of other malignancies except:

  * Malignancy treated with curative intent and with no known active disease present and felt to be at low risk for recurrence by treating physician. Current adjuvant hormonal therapy for disease treated with curative intent is permissible.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated carcinoma in situ without evidence of disease.
  * Low-risk prostate cancer on active surveillance
* Participants who are receiving any other investigational agents.
* History of severe allergic reactions attributed to compounds of similar chemical or biologic composition to obinutuzumab, venetoclax, or acalabrutinib. Patients with reactions to other CD20 monoclonal antibodies (e.g. rituximab, ofatumumab) are not excluded.
* Unable to receive prophylactic treatment for pneumocystis, herpes simplex virus (HSV), and herpes zoster (VZV) at start of treatment
* Known or suspected Richter's transformation or known CNS involvement
* Concurrent systemic immunosuppressant therapy (e.g., cyclosporine A, tacrolimus, etc., within 28 days of the first dose of study drug or chronic administration of >20 mg/day of prednisone within 7 days of the first dose)
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug.
* Ongoing or recent infection requiring intravenous antimicrobials at time of screening.
* Known bleeding disorders (e.g. von Willebrand's disease) or hemophilia.
* Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before screening.
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
* Major surgery within 4 weeks of first dose of study drug. If a subject had major surgery greater than 4 weeks prior to the first dose, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization.
* Baseline QTcF >480 ms. NOTE: This criterion does not apply to patients with a left bundle branch block.
* Patients who require warfarin or other vitamin K antagonists for anticoagulation (other anticoagulants are allowed).
* Patients who require treatment with proton pump inhibitors (see Appendix F). Subjects receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment on this study.
* Patients who require concurrent treatment with strong CYP3A inhibitors or strong CYP3A inducers are excluded from the study. If patients are receiving strong CYP3A inhibitors/inducers at time of screening but do not require continuous administration of these agents, these patients are eligible if there is a 3-day washout period between discontinuation of the strong CYP3A inhibitor/inducer and initiation of the first study drug, acalabrutinib.
* Patients who require concurrent treatment with P-gp inhibitors or narrow therapeutic index P-gp substrates are excluded from the study. If patients are receiving P-gp inhibitors or narrow therapeutic index P-gp substrates at time of screening but do not require continuous administration of these agents, these patients are eligible if there is a 3-day washout period between discontinuation of the P-gp inhibitor and initiation of acalabrutinib.
* Unable to swallow capsules or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel if thought by the investigator to compromise systemic absorption, active, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction.
* Patients with human immunodeficiency virus (HIV) or active hepatitis C virus (HCV) or hepatitis B virus (HBV) infection.
* Significant co-morbid condition or disease which in the judgment of the Principal Investigator would place the patient at undue risk or interfere with the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, compromise the subject's safety, or put the study outcomes at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2027-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew S. Davids, MD, MMSc, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Lifespan Cancer Institute, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davids MS, Ryan CE, Lampson BL, Ren Y, Tyekucheva S, Fernandes SM, Crombie JL, Kim AI, Weinstock M, Montegaard J, Walker HA, Greenman C, Patterson V, Jacobson CA, LaCasce AS, Armand P, Fisher DC, Lo S, Olszewski AJ, Arnason JE, Ahn IE, Brown JR. Phase II Study of Acalabrutinib, Venetoclax, and Obinutuzumab in a Treatment-Naive Chronic Lymphocytic Leukemia Population Enriched for High-Risk Disease. J Clin Oncol. 2025 Mar;43(7):788-799. doi: 10.1200/JCO-24-02503. Epub 2024 Dec 7. PMID 39645236
- [Derived] Davids MS, Lampson BL, Tyekucheva S, Wang Z, Lowney JC, Pazienza S, Montegaard J, Patterson V, Weinstock M, Crombie JL, Ng SY, Kim AI, Jacobson CA, LaCasce AS, Armand P, Arnason JE, Fisher DC, Brown JR. Acalabrutinib, venetoclax, and obinutuzumab as frontline treatment for chronic lymphocytic leukaemia: a single-arm, open-label, phase 2 study. Lancet Oncol. 2021 Oct;22(10):1391-1402. doi: 10.1016/S1470-2045(21)00455-1. Epub 2021 Sep 14. PMID 34534514

RESULTS

PARTICIPANT FLOW:
Groups:
- Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With Non-high-risk CLL Disease: * Acalabrutinib will be administered orally twice daily at 100 mg bid
  * Venetoclax will be administered orally once daily, with dose ramp-up from 20 mg up to a final dose of 400 mg
  * Obinutuzumab will be administered as per standard of care for 6 months with dosing at 100 mg on cycle 1 day 1, 900 mg on cycle 1 day 2, and then 1,000 mg on cycle 1 days 8, 15, and day 1 of cycles 2-6
  Venetoclax: Venetoclax is an oral drug that blocks the function of a protein called BCL-2. CLL cancer cells are thought to depend on the BCL-2 protein for their survival. By blocking BCL-2, venetoclax may kill cancer cells or stop them from growing.
  Obinutuzumab: Obinutuzumab is a type of drug called a monoclonal antibody. It targets a protein CD20 on the surface of the CLL cell, causing it to die
  Acalabrutinib: Acalabrutinib is a type of drug called a kinase inhibitor. It blocks a type of protein called Bruton Tyrosine Kinase (BTK) that helps CLL cells live and grow
- Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With High-risk CLL Disease: * Acalabrutinib will be administered orally twice daily at 100 mg bid
  * Venetoclax will be administered orally once daily, with dose ramp-up from 20 mg up to a final dose of 400 mg
  * Obinutuzumab will be administered as per standard of care for 6 months with dosing at 100 mg on cycle 1 day 1, 900 mg on cycle 1 day 2, and then 1,000 mg on cycle 1 days 8, 15, and day 1 of cycles 2-6.
  High-risk CLL disease (cohort 2), defined as 17p deletion and/or TP53 mutation
  Venetoclax: Venetoclax is an oral drug that blocks the function of a protein called BCL-2. CLL cancer cells are thought to depend on the BCL-2 protein for their survival. By blocking BCL-2, venetoclax may kill cancer cells or stop them from growing.
  Obinutuzumab: Obinutuzumab is a type of drug called a monoclonal antibody. It targets a protein CD20 on the surface of the CLL cell, causing it to die
  Acalabrutinib: Acalabrutinib is a type of drug called a kinase inhibitor. It blocks a type of protein called Bruton Tyrosine Kinase (BTK) that helps CLL cells live and grow
Period: Overall Study
Arm/Group | Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With Non-high-risk CLL Disease | Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With High-risk CLL Disease
Started | 37 | 35
Completed | 33 | 30
Not Completed | 4 | 5
Not completed — Death | 0 | 3
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Progressive Disease | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With Non-high-risk CLL Disease | Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With High-risk CLL Disease | Total
Number analyzed (Participants) | 37 | 35 | 72
Age, Continuous [Median (Full Range); unit: years] | 63 [41 to 78] | 65 [36 to 80] | 63 [36 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 27 | 22 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 35 | 34 | 69
  Other | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Rate of Bone Marrow (BM) Minimal Residual Disease (MRD) Negative Complete Response (CR) After 15 Cycles
Description: The rate of BM MRD was defined as the proportion of participants achieving CR and negative MRD based on 2018 IW-CLL criteria.
Time Frame: BM biopsy evaluated at baseline, cycle 4, 8, 16 on day 1. Relative to this endpoint is after 15 cycles
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With Non-high-risk CLL Disease | Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With High-risk CLL Disease
Number analyzed (Participants) | 37 | 35
proportion of participants | 0.378 [0.224 to 0.552] | 0.457 [0.283 to 0.638]

2. Secondary Outcome: Rate of Partial Response (PRR) After 15 Cycles
Description: The PRR was defined as the proportion of participants achieving PR based on 2018 IW-CLL criteria.
Time Frame: BM biopsy evaluated at baseline, cycle 4, 8, 16 on day 1. Relative to this endpoint is after 15 cycles
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With Non-high-risk CLL Disease | Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With High-risk CLL Disease
Number analyzed (Participants) | 37 | 35
proportion of participants | 0.54 [0.37 to 0.698] | 0.4 [0.236 to 0.582]

3. Secondary Outcome: Rate of Complete Response ( Including With Incomplete Count Recovery (CRi))
Description: The CR+CRi rate was defined as the proportion of participants achieving CR+CRi based on 2018 IW-CLL criteria.
Time Frame: BM biopsy evaluated at baseline, cycle 4, 8, 16, 25 on day 1.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With Non-high-risk CLL Disease | Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With High-risk CLL Disease
Number analyzed (Participants) | 37 | 35
proportion of participants
  After cycle 8 | 0.24 [0.12 to 0.41] | 0.2 [0.08 to 0.37]
  After cycle 16 | 0.432 [0.267 to 0.609] | 0.51 [0.336 to 0.689]
  After cycle 25 | 0.46 [0.29 to 0.63] | 0.62 [0.44 to 0.79]

4. Secondary Outcome: Median Progression-Free Survival (PFS)
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration between starting study therapy and documented disease progression (PD) or death, censored at time of last disease assessment.
Time Frame: Disease evaluated at baseline, cycle 4, 8, 16 on day 1, and every 3 months thereafter. Median follow-up for all patients was 55.23 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With Non-high-risk CLL Disease | Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With High-risk CLL Disease
Number analyzed (Participants) | 37 | 35
months | NA [NA to NA] — Median and bound of PFS not reached using KM method | 49.38 [49.38 to NA] — Upper bound of PFS not reached using KM method

5. Secondary Outcome: Median Overall Survival (OS)
Description: Overall Survival (OS) based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With Non-high-risk CLL Disease | Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With High-risk CLL Disease
Number analyzed (Participants) | 37 | 35
months | NA [NA to NA] — OS median and bounds not reached using KM method | NA [NA to NA] — OS median and bounds not reached using KM method

6. Secondary Outcome: Rate of Peripheral Blood (PB) MRD
Description: The rate of PB MRD was defined as the proportion of participants achieving negative MRD based on 2018 IW-CLL criteria. PB MRD evaluate by flow cytometry.
Time Frame: PB MRD evaluated on cycle 4, 8, 13, 16, 19, 22, 25, and every 3 cycles thereafter on day 1.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With Non-high-risk CLL Disease | Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With High-risk CLL Disease
Number analyzed (Participants) | 37 | 35
proportion of participants
  after 8 cycles | 0.68 [0.5 to 0.82] | 0.69 [0.51 to 0.83]
  after 16 cycles | 0.86 [0.71 to 0.95] | 0.8 [0.63 to 0.92]
  after 25 cycles | 0.89 [0.75 to 0.97] | 0.69 [0.5 to 0.84]

7. Secondary Outcome: Median Time to BM MRD-positive Disease Recurrence
Description: Median Time to BM MRD-positive Disease Recurrence based on the Kaplan-Meier method, is defined as the duration from the date of achieving MRD-negative status in the bone marrow to the date of first documented MRD-positive recurrence in the bone marrow, or death, whichever occurs first.
Time Frame: Disease evaluated at baseline, cycle 4, 8, 16 on day 1.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With Non-high-risk CLL Disease | Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With High-risk CLL Disease
Number analyzed (Participants) | 37 | 35
years | NA [NA to NA] — Time of median and bounds cannot be reached using KM method | NA [NA to NA] — Time of median and bounds cannot be reached using KM method

ADVERSE EVENTS:
Time Frame: AE collection thought entire study, on cycle 1 day 1, cycle 2 day 1, 2, 8, 15, 22, cycle 3 day 1 and 15, cycle 4 day 1, 2, 3, 8, 9, 15, 16, 22, 23, cycle 5 day 1 and 15, then day 1 on each cycle. Median duration of treatment is 25.56 months with range (0.56, 52.2).
Arm/Group | Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With Non-high-risk CLL Disease | Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With High-risk CLL Disease
All-Cause Mortality (participants affected / at risk) | 0/37 | 3/35
Serious Adverse Events (participants affected / at risk) | 10/37 | 9/35
Other Adverse Events (participants affected / at risk) | 37/37 | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With Non-high-risk CLL Disease (N=37) | Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With High-risk CLL Disease (N=35)
Colitis (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 2 | 2
Upper respiratory infection (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 | 1
Cardiac troponin I increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 3 | 0
Platelet count decreased (Investigations) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With Non-high-risk CLL Disease (N=37) | Acalabrutinib/Venetoclax/Obinutuzumab (AVO) With High-risk CLL Disease (N=35)
Anemia (Blood and lymphatic system disorders) | 23 | 14
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 2
Hemolysis (Blood and lymphatic system disorders) | 1 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 2
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 2
Chest pain - cardiac (Cardiac disorders) | 2 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 7 | 6
Sinus bradycardia (Cardiac disorders) | 0 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 4
Vertigo (Ear and labyrinth disorders) | 2 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 2 | 2
Blurred vision (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 2
Eye disorders - Other, specify (Eye disorders) | 1 | 3
Floaters (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Retinal vascular disorder (Eye disorders) | 0 | 1
Vision decreased (Eye disorders) | 2 | 0
Vitreous hemorrhage (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 10 | 7
Bloating (Gastrointestinal disorders) | 4 | 3
Constipation (Gastrointestinal disorders) | 7 | 9
Diarrhea (Gastrointestinal disorders) | 16 | 18
Dry mouth (Gastrointestinal disorders) | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 8
Dysphagia (Gastrointestinal disorders) | 0 | 1
Fecal incontinence (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 14 | 9
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Lip pain (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 20 | 17
Oral dysesthesia (Gastrointestinal disorders) | 3 | 0
Stomach pain (Gastrointestinal disorders) | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 5 | 6
Chills (General disorders) | 4 | 4
Edema face (General disorders) | 1 | 1
Edema limbs (General disorders) | 3 | 9
Edema trunk (General disorders) | 1 | 0
Facial pain (General disorders) | 1 | 0
Fatigue (General disorders) | 34 | 25
Fever (General disorders) | 6 | 7
Flu like symptoms (General disorders) | 0 | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 0
Generalized edema (General disorders) | 0 | 2
Localized edema (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 2 | 3
Pain (General disorders) | 4 | 8
Allergic reaction (Immune system disorders) | 0 | 1
Immune system disorders - Other, specify (Immune system disorders) | 0 | 2
Bacteremia (Infections and infestations) | 1 | 0
Bronchial infection (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1
Eye infection (Infections and infestations) | 0 | 2
Herpes simplex reactivation (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 4
Lip infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 3 | 3
Mucosal infection (Infections and infestations) | 0 | 1
Nail infection (Infections and infestations) | 0 | 2
Otitis externa (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Phlebitis infective (Infections and infestations) | 1 | 0
Shingles (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 6 | 5
Skin infection (Infections and infestations) | 2 | 2
Thrush (Infections and infestations) | 2 | 1
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 11 | 15
Urinary tract infection (Infections and infestations) | 1 | 4
Vaginal infection (Infections and infestations) | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 27 | 20
Fall (Injury, poisoning and procedural complications) | 2 | 5
Fracture (Injury, poisoning and procedural complications) | 1 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 8 | 9
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 3 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 6 | 13
Alkaline phosphatase increased (Investigations) | 4 | 11
Aspartate aminotransferase increased (Investigations) | 8 | 7
Blood bilirubin increased (Investigations) | 6 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 2
Creatinine increased (Investigations) | 12 | 10
Investigations - Other, specify (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1
Lymphocyte count increased (Investigations) | 2 | 1
Neutrophil count decreased (Investigations) | 29 | 18
Platelet count decreased (Investigations) | 28 | 20
Weight gain (Investigations) | 0 | 1
Weight loss (Investigations) | 1 | 2
White blood cell decreased (Investigations) | 7 | 1
Anorexia (Metabolism and nutrition disorders) | 5 | 7
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 8 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 6 | 3
Hyperlipidemia (Metabolism and nutrition disorders) | 1 | 2
Hypernatremia (Metabolism and nutrition disorders) | 4 | 0
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 | 6
Hyperuricemia (Metabolism and nutrition disorders) | 7 | 8
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 12 | 19
Hypokalemia (Metabolism and nutrition disorders) | 0 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 3
Hyponatremia (Metabolism and nutrition disorders) | 6 | 11
Hypophosphatemia (Metabolism and nutrition disorders) | 9 | 12
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 11
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 6 | 9
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 7
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Concentration impairment (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 7 | 11
Dysgeusia (Nervous system disorders) | 3 | 2
Dysphasia (Nervous system disorders) | 1 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 4
Facial muscle weakness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 28 | 26
Memory impairment (Nervous system disorders) | 1 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 2
Neuralgia (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 6
Presyncope (Nervous system disorders) | 0 | 2
Radiculitis (Nervous system disorders) | 0 | 1
Transient ischemic attacks (Nervous system disorders) | 1 | 1
Tremor (Nervous system disorders) | 2 | 0
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 6
Depression (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 6 | 8
Libido decreased (Psychiatric disorders) | 1 | 0
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 4
Hematuria (Renal and urinary disorders) | 2 | 3
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 | 1
Urinary frequency (Renal and urinary disorders) | 2 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 2
Urinary tract pain (Renal and urinary disorders) | 0 | 1
Urinary urgency (Renal and urinary disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Genital edema (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 2 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 4
Hair color changes (Skin and subcutaneous tissue disorders) | 1 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 10
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 7
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 15 | 3
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 1
Hematoma (Vascular disorders) | 1 | 0
Hot flashes (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 5 | 17
Hypotension (Vascular disorders) | 1 | 1
Thromboembolic event (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT03580928/Prot_SAP_001.pdf